CLINICAL TRIAL: NCT01392196
Title: Renal Denervation in Patients With Chronic Heart Failure & Renal Impairment
Brief Title: Renal Denervation in Patients With Chronic Heart Failure & Renal Impairment Clinical Trial
Acronym: SymplicityHF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No evidence of a physiological response; no significant safety concerns; post 24-month follow-up; Data Monitoring Committee agreed
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP085
Record Dates: First submitted 2011-07-07; First posted 2011-07-12 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Heart Failure
Keywords: Renal Impairment
MeSH Terms: conditions — Heart Failure; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Other): Renal Denervation
  Interventions: Procedure: Renal Denervation

INTERVENTIONS:
Procedure: Renal Denervation — Renal Denervation using the Symplicity Catheter in Heart Failure Population

SUMMARY:
This is a feasibility study enrolling up to 40 patients in Australia and Europe. The primary aim of the study is to demonstrate the renal denervation with the Symplicity Catheter is safe and determine the evidence of a response to renal denervation in patients with Heart Failure.

ELIGIBILITY:
Inclusion Criteria:

* Heart Failure patients NYHA Class II or III
* Renal Impairment Left Ventricular Ejection Function <40%
* GFR 30 to 75 mL/min/1.73m2
* Optimal stable medical therapy

Exclusion Criteria:

* Renal artery anatomy must be eligible for treatment as determined by Angiography, and
* History of prior renal artery intervention
* Single functioning kidney.
* Myocardial Infarction, unstable angina pectoris or cerebrovascular Accident within 3 months
* Systolic BP < 90 mmHG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-10; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Safety of Renal Denervation in Heart Failure patients as measured by Adverse Events | 6 month

SECONDARY OUTCOMES:
Ventricular function as measured by Echocardiography | 6 month
Renal function as measured by Glomerular Filtration Rate (GFR) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Henry Krum, MD, Principal Investigator — The Alfred
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia